CLINICAL TRIAL: NCT05903053
Title: Pilot Study: A Telehealth Intervention for Caregivers of Infants With Early Signs of ADHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003351
Record Dates: First submitted 2023-03-06; First posted 2023-06-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Infant Behavior; Infant Development; Self-Control; Self-Regulation, Emotion
MeSH Terms: conditions — Infant Behavior; Self-Control; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth Intervention (Experimental): A multiple baseline design across subjects will be used with varying introduction of treatment elements. Baseline periods will be 3, 5, and 7 sessions with the baseline period of 3 and 5 sessions repeated twice for subsequent participants. An intense intervention phase will follow the baseline phase in which 45-60 minute treatment sessions will occur twice per week over the course of 4-6 weeks for a total of 8 sessions. Each week during the intense intervention phase, caregiver coaches will introduce a new treatment technique to the caregiver and allow for caregiver practice with immediate feedback. At the conclusion of the intense intervention phase, coaches will provide "booster" sessions with the caregivers once weekly for 1 month (4 sessions total).
  Interventions: Behavioral: Early Self-Regulation Intervention

INTERVENTIONS:
Behavioral: Early Self-Regulation Intervention — Participants enrolled in a separate protocol (UC Davis IRB ID#1077801) will be invited to participate upon meeting eligibility criteria. All participants will receive the intake and exit assessment battery, with the intake assessment battery being completed as part of IRBNet ID#1077801. A multiple baseline design across participants will be used with varying introduction of treatment elements for a subset of enrolled intervention participants. An intense intervention phase will follow the baseline phase in which 45-60 minute intervention sessions will occur two times per week for approximately 4-6 weeks for a total of 8 sessions. At the conclusion of the intense intervention phase, coaches will provide "booster" sessions once weekly for a month (4 sessions total).

SUMMARY:
This project will build on the investigators' work focused on early identification of ADHD, expanding to the development of a feasibility/pilot intervention involving early intervention for such infants. The investigators will evaluate the effectiveness of a telehealth-delivered, caregiver-implemented supportive intervention for infants/toddlers show early self-regulation difficulties.

DETAILED DESCRIPTION:
This project will build on the investigators' work focused on early identification of ADHD, expanding to the development of a feasibility/pilot intervention involving early intervention for such infants. The investigators will evaluate the effectiveness of a telehealth-delivered, caregiver-implemented supportive intervention for infants/toddlers show early self-regulation difficulties.

Primary aims of this study include:

1. Develop and test a telehealth-delivered, parent-mediated intervention targeting infant/toddler self-regulation in natural contexts, to aid both infant and caregiver learning.
2. Identify, develop, and test measures/observations that can be gathered via telehealth contacts to assess ongoing change in infant and caregiver behavior over the course of the study.
3. Test acceptability and satisfaction of the intervention and the telehealth delivery for families receiving the intervention.

ELIGIBILITY:
Inclusion Critera:

Infants must be enrolled in UC Davis IRB protocol #1077801 and

* Be between the ages of 12-18 months at the time of intake assessment,
* Have a first-degree relative with ADHD (parent or sibling),
* Exhibit early symptoms of ADHD based on examiner observation as indicated by at least 1 subscale on the Behavior Rating Inventory for Children (BRIC) rated 4 or higher,
* Expression of at least 1 concern about the child's behavior/development by the caregiver.

Caregivers must:

* Be identified as the infants' primary caregivers,
* Be English-speaking,
* Have access to wired or wireless network technology to access the internet in their homes.

Exclusion Criteria:

* Birth before 33 weeks' gestation,
* Known genetic disorders (e.g., fragile X syndrome, Tuberous Sclerosis),
* History of traumatic brain injury,
* Severe visual, hearing, or motor impairment or fragile health condition that would prevent the child from validly participating in the assessment procedures, and
* A caregiver may be excluded from participation if the caregiver is already engaging in the majority of all possible caregiver treatment target behaviors at therapeutic levels during intake (Fidelity of Implementation scores of 80% or higher on each caregiver target behavior).

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Child attention regulation | Change from baseline at intervention session #8 (end of week 4)
  Child duration of orienting during the intervention sessions will be coded from video using a standardized behavioral coding paradigms developed within the investigators' lab.
Child inhibitory control | Change from baseline at intervention session #8 (end of week 4)
  Child frequency of grabbing behavior during the intervention sessions will be coded from video using a standardized behavioral coding paradigms developed within the investigators' lab.
Child emotion regulation | Change from baseline at intervention session #8 (end of week 4)
  Child frequency of negative affect during the intervention sessions will be coded from video using a standardized behavioral coding paradigms from the Lab-TAB. Higher levels equate to more negative affect.
Caregiver Fidelity of Implementation | Change from baseline at intervention session #8 (end of week 4)
  Caregiver fidelity of implementation (FI) of the intervention will be coded from 3-minute caregiver-child dyad intervention video probes to determine caregivers' FI of intervention techniques over the course of the study. This involves having experts in the intervention rate caregiver use of each of the intervention strategies on a 1-5 Likert rating scale, with a code of "1" meaning the caregiver did not implement the technique throughout the session and a code of "5" meaning the caregiver implemented the technique correctly throughout the session. An FI score of 80% (determined by total caregiver points out of the maximum possible points multiplied by 100) or higher for the entire intervention session indicates success in caregivers' FI of intervention techniques. Higher values represent greater fidelity.
Parent Satisfaction Rating | Immediately following session #8 (end of week 4)
  This is a measure of social validity, or acceptability, of the experimental treatment, to caregivers. This tool allows caregivers to rate the ease of implementation in the home and their opinions concerning treatment utility. Higher scores indicate greater satisfaction with the intervention.
Working Alliance Scale for Interventions with Children | Immediately following session #8 (end of week 4)
  This will be used to describe the response of the families to the intervention in terms of perceived alliance with the coach. Higher scores equate to more positive working alliance.
Lab-TAB Toy Retraction Task | Change from baseline at intervention session #8 (end of week 4)
  This task involves a standardized press for negative affect. The duration of negative affect during the task will be coded from video. Higher levels equate to more negative affect.

SECONDARY OUTCOMES:
Parent concerns interview | Change from baseline at intervention session #8 (end of week 4)
  The total number of parent concerns about child behavior and development will be examined. Fewer concerns reflects more positive outcomes.
Infant/Early Childhood Behavior Questionnaire (IBQ/ECBQ) - Effortful control | Change from baseline at intervention session #8 (end of week 4)
  The effortful control composite scores derived from these temperament rating scales will be examined. Higher scores reflect greater effortful control (i.e., more positive outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Miller, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No